CLINICAL TRIAL: NCT05388695
Title: To Observe the Long-term Efficacy and Safety of Dual-target Chimeric Antigen Receptor T Cells in the Treatment of Refractory Relapsed B Cell Hematologic Tumors
Brief Title: To Observe the Dual-target Chimeric Antigen Receptor T Cells in the Treatment of B Cell Hematologic Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Collaborators: Hebei Taihe Chunyu Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19+22 for B-ALL/NHL
Record Dates: First submitted 2022-05-19; First posted 2022-05-24 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: 19 and 22+ B Cell Hematologic Tumors; 19 and 20+ B Cell Hematologic Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 19+22 CART and 19+20 CART (Experimental): Eligible patients will be treated with 19+22 CAR-T and 19+20 CAR-T.
  Interventions: Biological: Autologous CD19/CD22/CD20 Chimeric Antigen Receptor T-cells

INTERVENTIONS:
Biological: Autologous CD19/CD22/CD20 Chimeric Antigen Receptor T-cells — Single or sequential injection of CD19, CD20 and CD22 CAR T cells.

SUMMARY:
To observe the long-term efficacy and safety of dual-target chimeric antigen receptor T cells in the treatment of refractory relapsed B cell hematologic tumors (at least 2 years).

DETAILED DESCRIPTION:
This study is open single-arm prospective clinical study To relapse/refractory blood B cell tumor patients as the subjects, according to the expression of tumor cells, gives the corresponding double targets CART cell injection treatment, follow-up observation of the adverse reactions and the treatment effect of the drug to the data (at least 2 years), assessment of double targets CAR - T Long-term efficacy and safety of cell injection

ELIGIBILITY:
Inclusion Criteria:

1. Refractory and relapsed B-cell tumor determined by clinical diagnosis, B cell tumors include the following three categories: B cell acute lymphocyte leucocyte; Inert B cell lymphoma (CLL、 FL、 MZL); Aggressive B-cell lymphoma (DLBCL、 BL、 MCL);
2. CD19 positive and CD20 positive or CD22 positive were detected by immunohistochemistry or flow cytometry; 3.18 years old≤age≤70 years old;

4.Estimated survival time>3 months; 5.ECOG Scores: 0~2; 6.There should be at least one measurable tumor foci according to RECIST Version 1.1; 7.The functions of vital organs must meet the following conditions: EF>50%, and no obvious abnormality of electrocardiogram; SpO2≥92%; Cr≤1.5ULN; ALTand AST≤5ULN, TBil≤3ULN; 8.Subjects planning to become pregnant must agree to use contraception prior to enrolling in the study and after six months of study duration; inform the investigator immediately if the subject becomes pregnant or suspects pregnancy; 9.The subject or guardian understands and signs the informed consent.

Exclusion Criteria:

1. With other diseases that are not effectively controlled, including, but not limited to, persistent or poorly controlled infections symptomatic congestive heart failure unstable angina arrhythmia poorly controlled pulmonary disease or psychiatric disease;
2. Presence of other malignant tumors;
3. There are severe infections that cannot be effectively controlled;
4. Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive, peripheral blood hepatitis B virus (HBV)DNA higher than the detection limit should be excluded; If hepatitis C virus (HCV) antibody positive, peripheral blood HCV RNA positive need to exclude; Cytomegalovirus (CMV)DNA positive; Epstein-barr virus DNA positive in peripheral blood;
5. Known positive serology for human immunodeficiency virus (HIV) or syphilis;
6. A history of severe allergies to biological products (including antibiotics);
7. Patients with relapses after allogeneic hematopoietic stem cell transplantation with grade 3-4 acute graft-versus-host disease (GvHD);
8. Female patients who are under pregnancy and/or lactation;
9. Active autoimmune disease requiring systemic immunosuppressive therapy;
10. Conditions that the investigator believes may increase the risk to the subject or interfere with the results of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-04-08 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy: Remission Rate | Up to 3 months
  Remission Rate includes complete remission(CR)、CR with incomplete blood count recovery(CRi)、No remission(NR)

CONTACTS AND LOCATIONS:
Overall Officials: Jia Wei, PhD&MD, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] He S, Peng J, Yang X, Meng F, Huang L, Huang L, Tian W, Gao Z, Zhao J, Wang Z, Wei J. Peripheral Blood Smears Distinguish Infective Fever after CAR-T Therapy. Front Biosci (Landmark Ed). 2023 Nov 24;28(11):299. doi: 10.31083/j.fbl2811299. PMID 38062808